CLINICAL TRIAL: NCT00996671
Title: A Phase I, Randomized, Single-Blind, Placebo-Controlled Dose-Escalation Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Food Effect Following Single Oral Doses of the Focal Adhesion Kinase Inhibitor, GSK2256098, in Healthy Subjects
Brief Title: Phase I Study to Evaluate Safety, Pharmacokinetics and Pharmacodynamics of GSK2256098 in Healthy Volunteers
Acronym: FTIH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 113581
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Cancer
Keywords: focal adhesion kinase inhibitor; healthy volunteers; first time in human
MeSH Terms: conditions — Neoplasms | interventions — GSK2256098

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose Escalation Cohorts (Experimental): single dose administration escalating doses starting at 20 mg and continue escalation; the highest dose in this study will not exceed the mean Day 1 exposure in male dogs at the NOAEL dose (6 mg/kg/day).
  Interventions: Drug: GSK2256098; Drug: Placebo
- Food effect Cohort (Experimental): Dose to be selected based on emerging safety and PK data; subjects will be given FDA standard high fat meal followed by single dose of study drug.
  Interventions: Drug: GSK2256098

INTERVENTIONS:
Drug: GSK2256098 — focal adhesion kinase inhibitor given as a single dose
Drug: Placebo — Placebo to be used as comparator for GSK2256098
  Arms: Dose Escalation Cohorts

SUMMARY:
The purpose of this study is to test the safety of a new drug and to look at how the drug is handled by your body. This is the first time the drug will be given to people, the drug has been safely given to animals over many days at higher doses than will be given in the study. The study will be done in healthy men and woman to determine what effects, good or bad, it has on thier health. This study will find out:

If the drug has any side effects after one dose of the drug is given? How much of the drug gets into the bloodstream, and how long does the body take to get rid of it? If the drug causes any changes to a substance that is in skin, hair or blood.

DETAILED DESCRIPTION:
This study represents the first administration of the focal adhesion kinase (FAK) inhibitor GSK2256098 to humans to evaluate the safety, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary food effect following single oral doses in adult healthy subjects before proceeding to studies in subjects with cancer that will be given at higher doses over an extended period of time. FAK is a protein in the body that is important in cancer development. Objectives of the study will be to characterize the safety of single doses of GSK2256098; to characterize the single dose PK of GSK2256098 in the presence and absence of food; to examine the dose proportionality of GSK2256098 PK parameters following single dose administration; and to characterize the effect of single doses of GSK2256098 on phospho-FAK (pFAK) tyrosine 397 (Y397) levels in skin and hair follicles. Dose- and concentration-effect relationships for various safety parameters will be explored as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* AST, ALT, alkaline phosphatase and bilirubin less than or equal to 1.5 X ULN (isolated bilirubin >1.5 X ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%).
* Urine microalbumin: creatinine ratio < 300 mg/g.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory].
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until the end of the follow-up period.
* Body weight greater than or equal to 50 kg and body mass index (BMI) within the range 18.5 to 30.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Average QTcF < 450 msec (based on averaged results of three ECGs).

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within three months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of alcohol consumption within six months of the study defined as:

an average weekly intake of > 21 units for males or > 14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.

* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, five half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities or investigational products within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within seven days (or 14 days if the drug is a potential enzyme inducer) or five half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum hCG test at screening or positive urine hCG test prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Subjects who have asthma or a history of asthma or reactive airway disease.
* History of regular tobacco use or nicotine containing products within three months prior to screening or a positive urine cotinine test result indicative of smoking at screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or kumquats, pummelos, exotic citrus fruit (i.e., star fruit, bitter melon), grapefruit hybrids or fruit juices from seven days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-11-06 (Actual); Primary Completion 2010-03-17 (Actual); Study Completion 2010-03-17 (Actual)

PRIMARY OUTCOMES:
To characterize the safety of single doses of GSK2256098 in adult healthy subjects | within 10-14 days following administration of study drug
To characterize the single dose pharmacokinetics of GSK2256098 in blood and urine in adult healthy subjects | 14 days after administration of study drug

SECONDARY OUTCOMES:
To examine the dose proportionality of GSK2256098 pharmacokinetic parameters following single dose administration in healthy subjects | 14 days
To explore dose- and concentration-effect relationships for various safety parameters, if appropriate | 14 days
To estimate the effect of high fat/calorie meal on the pharmacokinetics, safety, and tolerability of a single dose of GSK2256098. | 14 days
To explore and potentially identify small molecules or cytokines in plasma which may serve as biomarkers for future studies | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 113581 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113581?search=study&search_terms=113581#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 113581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113581 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register